CLINICAL TRIAL: NCT02423733
Title: Can E-therapies Reduce Waiting Lists in Secondary Mental Health Care? A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Simon Hatcher, Vice Chair Research, Department of Psychiatry, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014001
Record Dates: First submitted 2015-04-13; First posted 2015-04-22 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Depression
Keywords: depression; dysthymia; cognitive behavioural therapy; CBT; problem-solving therapy; PST; waitlist; secondary mental health care; mental health; e-therapy; computerized therapy
MeSH Terms: conditions — Depression; Dysthymic Disorder; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): In addition to their usual clinical care will also be given written information about web sites that provide information on depression but will not be specifically directed to The Journal.
- Computerized Therapy (Experimental): In addition to their usual clinical care they will receive an invitation to use The Journal supported by an e-therapy coach who will provide patients with weekly email or telephone contact. The e-therapy coach will have a guideline script for each lesson of The Journal to reinforce the topic of each lesson, help identify and support patients in their goals and to coach them in goal setting and the techniques of problem solving.
  Interventions: Other: The Journal

INTERVENTIONS:
Other: The Journal — "The Journal" is a free internet based program for the self-management of depression (www.depression.org.nz) that was developed in New Zealand and capitalizes on the social marketing appeal of Sir John Kirwan, an ex All Black who has described his experiences of depression to help destigmatize mental illness. . The self-help program is based on the cognitive behavioral techniques of behavioral activation and problem solving which teaches patients the skills of problem solving and delivers an evidence based intervention which is personalized for their individual care.
  Arms: Computerized Therapy

SUMMARY:
Depression is common and disabling but access to specialist treatment is often delayed with waiting lists of up to a year not uncommon. Also treatment is frequently limited to drug therapies because of long waiting lists to see psychological therapists face to face despite recommendations by NICE (The National Institute for Health and Clinical Excellence) and others about the importance of non-drug therapies. One way to address this problem is to use computerized e-therapies which deliver structured cognitive behavioral treatment where the therapy can be accessed in a location and at a time that is convenient for patients and where there is no waiting list. Previous randomized controlled trials of e-therapies for depression have mainly been in people recruited through the internet or in clinical populations with mild disorders where many participants do not complete the on-line course. Despite this there is some evidence that clinician-assisted computerized cognitive behavior therapy can result in significant improvements in depression with reduced demands on clinician time. To date there have been no trials of clinician assisted e-therapy in secondary care.

Therefore the aim of this clinical trial is to answer the question "In patients on the waiting list for the mood program does a computerized therapy with an e-therapy coach compared to written information about depression and the availability of computerized treatments result in better outcomes, quicker improvements and the use of fewer resources after 12 weeks". The study will be a randomized controlled trial with health service use and PHQ-9 as the main outcome measures.

DETAILED DESCRIPTION:
Depression is common and disabling but the evidence is that fewer than half of people with depression seek any treatment and few receive any help from specialized mental health professionals (1). In secondary care treatment is often limited to drug therapies because of long waiting lists to see psychological therapists face to face despite recommendations by NICE and others about the importance of non-drug therapies (2). At The Royal Ottawa Health Care Group the waiting time to be seen in the Mood Program is between nine months and a year. One way to address this problem is to use computerized e-therapies which deliver structured cognitive behavioral treatment via a computer (3). The appeal of e-therapies is that they solve several problems. Firstly they are convenient for users. They can be used at any time and can be accessed in different locations. Secondly there is no waiting for appointments. Last for health providers they address the workforce issue of a lack of trained providers of effective interventions. If e-therapies can be shown to be acceptable, feasible and effective there is no reason why these computerized therapies could not replace humans leaving qualified professionals to focus on more complex management problems. This may lead to the development of new role which in this proposal is an e-therapy coach.

Previous randomized controlled trials of e-therapies for depression have mainly been in people recruited through the internet or in clinical populations with mild or "sub-clinical" disorders(4). The difficulty with these populations is that there is a high rate of spontaneous remission. However systematic reviews have consistently found a significant moderate effect of computerized therapies in reducing depressive symptoms compared to control conditions (5, 6). A further problem is that many people fail to complete the course of e-therapy (although this also applies to face to face therapies). There is a need for randomized controlled trials of e-therapies in clinical populations using novel techniques to maximize the dose of e-therapy without losing the potential health workforce benefits.

A potentially attractive solution is to enable clinician-assisted computerized cognitive behavior therapy. For this proposal the investigators plan to use an e-therapy coach who would coach people through the on-line therapy. In this model the clinician acts in the role of a coach to support the patient progress through the computerized treatment - the clinician does not need to deliver the non-drug therapy themselves. There is some evidence that this can result in significant improvements in depression with reduced demands on clinician time(7). However previous trials have been done using participants with relatively less severe depression who may not have seen clinicians as part of their usual care (8). Also the outcome measures are usually only self-rating scales rather than objective measures of function. To date there have been no trials of clinician assisted e-therapy in secondary care.

"The Journal" (9) a free internet based program for the self-management of depression (www.depression.org.nz) was developed in New Zealand and capitalizes on the social marketing appeal of Sir John Kirwan, an ex All Black who has described his experiences of depression to help destigmatize mental illness. However in Canada John Kirkan is unknown so one hypothesis the investigators will test in this study is whether the social marketing by a celebrity is necessary for the effective use of an e-therapy. The self-help program is based on the cognitive behavioral techniques of behavioral activation and problem solving which teaches patients the skills of problem solving and delivers an evidence based intervention which is personalized for their individual care. The problem solving approach was derived from a large randomized control trial of face to face problem solving used in people who presented to emergency departments with intentional self-harm (10).

Usage data from New Zealand shows that the depression.org web site was visited by 700,000 people in its first year (the population of New Zealand is 4.2 million) with 20,000 registered with The Journal and 13,000 active users. About 1500 people a month register to start the program with about three quarters of people recording significant improvement. Although the program was designed for depression of mild to moderate severity the evidence shows that nearly a third of people who access the program have more severe depression. The mean PHQ-9 score at the start of the program is 16 which reduces to 10 after 3 sessions and 7 by the end of the program. The change in depression scores is most marked for severe depression with only 5% of people scoring in the severe range at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older .
* Referred to the Youth, Geriatric, or Mood and Anxiety Psychiatry Programs at the Royal Ottawa Mental Health Centre for any depressive symptoms.
* Has been triaged to the Youth, Geriatric, or Mood and Anxiety Psychiatry Programs at the Royal Ottawa Mental Health Centre.

Exclusion Criteria:

* Is unable to read or write in English
* Has cognitive impairments that render participant unable to use a computer
* Does not have access to a computer
* Does not have an OHIP number

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Scores on PHQ-9 Scale | Baseline, 2, 6 and 12 weeks
  Measures severity of depressive symptoms.

SECONDARY OUTCOMES:
Change in Scores on SF-12 Scale | Baseline, 6 and 12 weeks
  A generic measure of function and well being
Change in Scores on EQ-5D Scale | Baseline, 6 and 12 weeks
  A generic health-related quality of life index that can be related to costs
Internet Use Questionnaire | 12 weeks
  Record of internet resources used relating to health concerns assessed by self-report
Time Off Work Questionnaire | 12 weeks
  To assess cost of treatment
Hospital Admission from ICES data | 12 weeks
  To assess cost of treatment
Outpatient appointments from ICES data | 12 weeks
  To assess cost of treatment
Medication use from ICES data | 12 weeks
  To assess cost of treatment

OTHER OUTCOMES:
Demographic Questionnaire | Baseline
  To describe similarities and differences between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Simon Hatcher, MD., Principal Investigator — University of Ottawa
Locations (1):
- Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Andrews G, Titov N. Depression is very disabling. Lancet. 2007 Sep 8;370(9590):808-9. doi: 10.1016/S0140-6736(07)61393-2. No abstract available. PMID 17826154
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] So M, Yamaguchi S, Hashimoto S, Sado M, Furukawa TA, McCrone P. Is computerised CBT really helpful for adult depression?-A meta-analytic re-evaluation of CCBT for adult depression in terms of clinical implementation and methodological validity. BMC Psychiatry. 2013 Apr 15;13:113. doi: 10.1186/1471-244X-13-113. PMID 23587347
- [Background] Titov N, Andrews G, Davies M, McIntyre K, Robinson E, Solley K. Internet treatment for depression: a randomized controlled trial comparing clinician vs. technician assistance. PLoS One. 2010 Jun 8;5(6):e10939. doi: 10.1371/journal.pone.0010939. PMID 20544030
- [Background] Hatcher S, Sharon C, Parag V, Collins N. Problem-solving therapy for people who present to hospital with self-harm: Zelen randomised controlled trial. Br J Psychiatry. 2011 Oct;199(4):310-6. doi: 10.1192/bjp.bp.110.090126. Epub 2011 Aug 4. PMID 21816868
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Depression: Evidence Update April 2012: A summary of selected new evidence relevant to NICE clinical guideline 90 'The treatment and management of depression in adults' (2009) [Internet]. London: National Institute for Health and Clinical Excellence (NICE); 2012. No abstract available. Available from http://www.ncbi.nlm.nih.gov/books/NBK552056/ PMID 31886986
- [Background] Marks I, Cavanagh K, Gega L. Hands-on help: Computer-aided psychotherapy. Psychology Press Taylor and Francis, 2007
- [Background] Cowpertwait L, Clarke D. Effectiveness of web-based psychological interventions for depression: A meta analysis. International Journal of Mental Health and Addiction. 2013; 11: 247-68
- [Background] Vernmark K, Lenndin J, Bjarehed J, Carlsson M, Karlsson J, Oberg J, Carlbring P, Eriksson T, Andersson G. Internet administered guided self-help versus individualized e-mail therapy: A randomized trial of two versions of CBT for major depression. Behav Res Ther. 2010 May;48(5):368-76. doi: 10.1016/j.brat.2010.01.005. Epub 2010 Feb 2. PMID 20152960
- [Background] Ministry of Health. 2009. www.depression.org.nz.
- [Derived] MacLean S, Corsi DJ, Litchfield S, Kucharski J, Genise K, Selaman Z, Testa V, Hatcher S. Coach-Facilitated Web-Based Therapy Compared With Information About Web-Based Resources in Patients Referred to Secondary Mental Health Care for Depression: Randomized Controlled Trial. J Med Internet Res. 2020 Jun 9;22(6):e15001. doi: 10.2196/15001. PMID 32515740